CLINICAL TRIAL: NCT00000430
Title: Clinical Trial of Continuous Low-Dose Hormone Replacement Therapy Combined With Alendronate in Postmenopausal Women With Low Bone Density
Brief Title: Low-Dose Hormone Replacement Therapy and Alendronate for Osteoporosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01 AR92237; NIAMS-040
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2004-02

CONDITIONS: Osteopenia; Osteoporosis
Keywords: Osteoporosis; Osteopenia; Postmenopausal women; Hormone replacement therapy; Alendronate
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Alendronate; Estrogens

INTERVENTIONS:
Drug: Alendronate
Drug: Estrogen/progestin therapy

SUMMARY:
Osteoporosis, a condition in which bones are fragile and break easily, is a major health problem for postmenopausal women. Research studies have shown that both estrogen/progestin replacement therapy (hormone replacement therapy, or HRT) and alendronate are effective in preventing and treating osteoporosis. However, because these drugs work in somewhat different ways, a combination of the two drugs might protect women from osteoporosis better than either drug alone. In this study we will test whether HRT and alendronate given together for 3.5 years to postmenopausal women with low bone mass will have a greater effect on bone than either HRT or alendronate given alone. We will also give every participant in this study calcium and vitamin D supplements.

DETAILED DESCRIPTION:
Clinical trials of estrogen/progestin replacement therapy (HRT) and a bisphosphonate, alendronate (ALN), have demonstrated that both are effective in causing gains in bone mass and preventing bone loss and fractures in postmenopausal women. The FDA has approved both these drugs for prevention and treatment of fractures, and both are widely used in clinical practice. Because both are approved and effective, and they work by different mechanisms, many patients and their physicians ask whether both should be taken in combination, particularly in cases of severe disease. The question is asked frequently because of the high incidence of osteoporosis among women and the need for long-term prevention and treatments that often last decades.

Indeed, physicians are using ALN and HRT together without adequate scientific support for the assumption that the combination is more effective than either given alone.

Clinical trials are now underway to test conventional doses of HRT given as conjugated equine estrogens (CEE), 0.625 mg/day or its equivalent, combined with ALN, 10 mg/day. However, researchers are not studying the bone-sparing effectiveness of the combined administration of ALN and low-dose continuous HRT given as CEE, 0.3 mg/d, along with medroxyprogesterone, 2.5 mg/d (MP). This low-dose continuous HRT regimen is attractive because of better convenience, better patient tolerance, and reduced risk of breast cancer and other safety concerns associated with conventional higher doses. Further, we have recently demonstrated that the bone-sparing effect of this regimen is comparable to that of higher doses.

The long-term objective of this study is to test the hypothesis that the combined therapy shows a greater bone effect than does either treatment given alone. Our specific aim is to conduct a 3.5 year, randomized, double-blind, controlled trial of low-dose, continuous HRT combined with alendronate, 10 mg/d (ALN), in three groups (72 people per group) of estrogen-deprived postmenopausal women over age 60. We will give Group 1 low-dose HRT, Group 2 ALN, and Group 3 both low-dose HRT and ALN. We will give calcium and vitamin D supplements to people in all three groups.

The primary outcome measures will be spine bone mineral density (SpBMD) and total hip bone mineral density (HipBMD) measured by dual energy X-ray absorptiometry (DXA). Secondary outcome measures will be total body bone mineral content and forearm bone mineral content. In addition, we will perform studies to characterize the mechanism of the effects of these regimens. These studies will consist of measurements of urinary bone resorption markers, serum bone formation markers, calcium excretion, calcium absorption, and application of a model developed in our laboratory to estimate and compare the magnitudes of the anabolic effects (if any) of all three interventions on SpBMD and HipBMD.

We have reported data showing that both agents have an anabolic effect on bone in humans, meaning that they cause an increase in bone mass beyond that explained by a remodeling transient brought about by reduction in bone remodeling rates. Further, research has shown that HRT and ALN affect bone by different mechanisms. Thus, this combination may have an additive effect on bone resulting in bone gain beyond that previously seen with other interventions. This project will provide much-needed information to physicians and their patients on the benefits and safety of this combination regimen so that they can make "evidence-based" decisions on the choice of interventions to prevent and treat osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 60 years of age.
* Good general health.
* Willingness to participate in this 3.5 year study.
* Ability to give informed consent.
* Ability to live independently and travel to the research center for visits (we will provide transportation on a limited basis).
* Spine bone mineral density (BMD) (L1-4) T-score between -1.0 and -2.5, or a hip T-score between -1.0 and -2.5. A T-score of -1.0 is equal to a bone mass of one standard deviation below the mean peak bone mass in healthy young adult women.

Exclusion Criteria:

* Any history of cancer except the following: (a) superficial basal or squamous cell carcinoma of the skin which has been completely resected or resolved by a topical chemotherapeutic agent, and (b) other malignancies treated curatively at least 10 years previously, without any evidence of recurrence.
* Abnormal transvaginal ultrasound that has not been investigated and cleared by endometrial biopsy.
* History of low-trauma hip or spine fracture previously diagnosed.
* Serious residuals from cerebral vascular disease.
* Diabetes mellitus, except for easily controlled, non-insulin dependent or insulin dependent diabetes mellitus without significant microvascular or neuropathic disease.
* Serum creatinine >1.9 mg/dl.
* Chronic liver disease or alcoholism.
* Treatment with bone active agents such as fluoride or bisphosphonates within the previous 2 years.
* Treatment with calcitonin, estrogen, or a selective estrogen receptor modulator within the previous 6 months.
* Systemic corticosteroid therapy at pharmacologic levels for more than 6 months duration.
* Any corticosteroid therapy within the previous 6 months.
* Treatment with anticonvulsant therapy within the previous year.
* Clinically significant abnormalities on pre-study laboratory or clinical screens.
* Treatment with thyroid hormone is accepted, provided the patient is euthyroid at the time of entry, and the serum TSH by ultrasensitive assay is normal.
* Uncontrolled hypertension.
* Unstable angina.
* Myocardial infarction within 1 year prior to entry.
* Evidence of metabolic bone disease, e.g. hyper- or hypoparathyroidism, Paget's disease, osteomalacia, osteogenesis imperfecta, or others.
* Active rheumatoid arthritis or collagen disease.
* Recent major gastrointestinal disease (within the past year) such as peptic ulcer, malabsorption, chronic ulcerative colitis, regional enteritis, or any significant chronic diarrhea state.
* Tobacco use at a level of more than 10 cigarettes per day.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 1999-10; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Robert R. Recker, MD, Principal Investigator — Creighton University Osteoporosis Research Center; Joan M. Lappe, PhD, RN, Study Director — Creighton University Osteoporosis Research Center
Locations (1):
- Creighton University Osteoporosis Research Center, Omaha, Nebraska, United States